CLINICAL TRIAL: NCT01541202
Title: A Phase III, Multi-center,Randomized, Double-blind, Based on Standard Therapy, Placebo-controlled Study of the Survival of Recombinant Human Neuregulin-1β in Patients With Chronic Systolic Heart Failure
Brief Title: Study of the Survival of Recombinant Human Neuregulin-1β in Chronic Heart Failure (CHF) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor has designed another study to replace the current study
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-305
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2012-02

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; neuregulin; mortality
MeSH Terms: conditions — Fibromatosis, Gingival, 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo in addition to standard therapy
  Interventions: Drug: Placebo
- rhNRG-1 (Experimental): rhNRG-1 in addition to standard therapy
  Interventions: Drug: rhNRG-1

INTERVENTIONS:
Drug: rhNRG-1 — 10 hours per day i.v drip for the first 10 days (0.6ug/kg/day), followed by weekly 10 minutes i.v bolus (0.8ug/kg/day), from the 3rd week for 23 weeks
  Arms: rhNRG-1
Drug: Placebo — 10 hours per day i.v drip for the first 10 days (0ug/kg/day), followed by weekly 10 minutes i.v bolus (0ug/kg/day), from the 3rd week for 23 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of rhNRG-1 in reducing the death rate of heart failure.

DETAILED DESCRIPTION:
The mortality of chronic heart failure patients remains high, in spite of current treatment. RhNRG-1(recombinant human neuregulin-1)directly work on the cardiomyocyte and restored the normal structure and function of it. Both the preclinical trial and phase II clinical trail have confirmed that rhNRG-1 effectively enhance the heart function, reverse the remodeling of left ventricular, and reduce all-cause mortality in heart failure animals and humans. In this phase III study, the investigators will further confirm the efficacy of rhNRG-1 in reducing the death rate of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75, both sex.
2. Left ventricular ejection fraction (LVEF)≤40% (ECHO).
3. NYNA functional class II OR III.
4. Diagnosed as chronic systolic heart failure (history, symptoms, signs), no in-hospital history in the last one month.
5. Receiving standard therapy for chronic heart failure, reach target dose or max tolerable dose for one month, or has not changed the dose for the last one month.
6. Capable of signing the informed consent form.

Exclusion Criteria:

1. new chronic heart failure patients, or patients receiving standard therapy on chronic heart failure for less than 3 months.
2. NYNA functional class I OR IV.
3. Patients with acute MI, hypertrophic cardiomyopathy, constrictive pericarditis, significant valvular pathological change or congenital heart diseases, primary or secondary severe pulmonary artery hypertension.
4. Ischemic heart failure without recanalization or with recanalization in recent six months.
5. acute MI in the last 3 months.
6. unstable angina.
7. Patients with acute pulmonary edema or acute hemodynamic disorder.
8. Chronic heart failure patients with acute hemodynamic disorder or acute decompensation in the last 1 month.
9. Patients with right heart failure caused by pulmonary disease.
10. Patients diagnosed with pericardial effusion or pleural effusion, or evidenced by B-type ultrasonic (>50ml).
11. Cardiac surgery or cerebrovascular accident within recent six months.
12. Preparing for heart transplantation or CRT, or has received CRT.
13. Serious ventricular arrhythmia (multi-morphological premature ventricular contraction more than 5 times/min, frequent paroxysmal ventricular tachycardia or triple rate).
14. Serious hepatic or renal dysfunction (Cr>2.0mg/dl, AST or ALT 5 times above the normal upper limit).
15. Serum potassium <3.2 mmol/L or >5.5 mmol/L.
16. Systolic blood pressure <90mmHg or >160mmHg.
17. Pregnant or plan to pregnant.
18. Patients who participated in any clinical trial in the recent three months.
19. Subject with a life expectancy less than 6 months as assessed by the investigator.
20. Serious nervous system diseases (Alzheimer's disease, advanced Parkinsonism),lower limb defects, or deaf-mute.
21. History of any malignancy or suffering from cancer,or biopsy proven pre-malignant condition (eg DICS or cervical atypia).
22. Evidence (physical examination,CXR,ECHO or other tests) shows some active malignancy or adenoidal hypertrophy or neoplasm has effect on heart function or endocrine system, eg pheochromocytoma or hyperthyroidism.
23. Judging by the investigator, the patients could not complete the study or adhere to the study requirements (due to the management reasons or others).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2012-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 1 year

SECONDARY OUTCOMES:
sudden death | 1 year
death caused by cardiovascular events | 1 year
rehospitalization | 1 year
hospitalization caused by worsening heart failure | 1 year
cardiac function | 1 year
NYHA functional classification | 1 year
6 minute walking distance | 1 year
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Ph.D, Principal Investigator — Cardiovascular Institute and Fuwai Hospital
Locations (46):
- China (46):
  - Beijing Anzhen Hospital, Affiliate of Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chao Yang Hospital, Affiliate of Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Xuanwu hospital of Capital Medical University, Beijing, Beijing Municipality
  - Cardiovascular Institute and Fuwai Hospital, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Xinqiao Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yet-Sen University, Guangzhou, Guangdong
  - Haikou Municipal Peoples Hospital, Haikou, Hainan
  - Bethune Peace Hospital, Shijiazhuang, Hebei
  - Teda International Cardiovascular Hospital, Tianjin, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First hospital affiliated to Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - The Second Hospital affiliated to Suzhou University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical School, Xuzhou, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Affiliate Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Hospital affiliated to Jilin University, Changchun, Jilin
  - The First Hospital affiliated to Dalian Medical University, Dalian, Liaoning
  - The first affiliated hospital of Liaoning medical college, Jinzhou, Liaoning
  - The First Hospital of China Medical College, Shengyang, Liaoning
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The first people's hospitial of Shanghai, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical College, Taiyuan, Shanxi
  - The second hospital of Xi'an jiaotong university, Xi’an, Shanxi
  - Huaxi Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Kunming General Hospital of Chengdu Military Region, Kunming, Yunnan
  - The Second Hospital of Kunming Medical College, Kunming, Yunnan
  - Sir Run Run Shaw Hospital affiliated to School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Hospital affiliated to School of Medicine, Zhejiang University, Hangzhou, Zhejiang